## CONSENT FORM FOR PARTICIPANTS IN RESEARCH PROJECTS





Title of project: An exploratory randomised control trial of a single session intervention combined with a socially assistive robot to promote emotion regulation competence in university students Ethical review reference number: 28406 Version number: March 2022 - v1.1 Tick or initial 1. I confirm that I have read and understood the information sheet dated March 2022 v1.1 for the above project. I have had the opportunity to consider the information and asked questions which have been answered to my satisfaction. 2. I consent voluntarily to be a participant in this project and understand that I can refuse to take part and can withdraw from the project at any time without giving any reason. And that if I withdraw consent up until 2 weeks after the last completed survey, any data I have provided to that point will be destroyed; that I can withdraw consent from the follow-up interview up to 1 week after it took place; and that I will not be able to withdraw my data from the focus group. 3. I consent to the processing of my personal information for the purposes explained to me in the Information Sheet. I understand that such information will be handled under the terms of UK data protection law, including the UK General Data Protection Regulation (UK GDPR) and the Data Protection Act 2018. 4. I understand that my information may be subject to review by responsible individuals from the College for monitoring and audit purposes. 5. I understand that confidentiality will be respected unless there are compelling and legitimate reasons for this to be breached, such as if any actions or planned actions are discovered that are likely to result in serious or immediate harm to me or others. Following their duty of care, the researchers will report to the relevant authorities (e.g. Counselling Services at Oxford University) any possible harm or danger to you or others. 6. I understand that whilst the research team will maintain confidentiality on any data collected, the research team is unable to guarantee confidentiality of the focus groups due to the chance of a focus group participant breaking confidentiality. 7. I understand that any information given by me (that is questionnaires data and quotes from interviews) may be used in future reports, academic articles, publications or presentations by the researchers of this project (including webpages), but my personal information will not be included and I will not be identifiable. 8. I agree that the research team may use my data for future research and understand that any such use of identifiable data would be reviewed and approved by a research ethics committee. (In such cases, as with this project, data would not be identifiable in any report). 9. I consent to be invited to take part in one online interview at the end of the Trinity Term 2022 to discuss my experience in the study. 10. I consent to be invited to take part in one online focus group at the end of the Trinity Term 2022 to discuss how the intervention could be improved for university students.

| And I agree to maintain the confidentiality of the focus group by not disclosing any confidential information with others. | | |
|---|---|---|
| 11. I consent to my participation in the interview and/or focus group being audio recorded. | | |
| 12. I consent to my participation in the interview and/or focus group being video recorded. | | |
| 13. I agree to my pseudo-anonymised data being shared with external collaborators outside the UK (i.e. project researchers at Stony Brook University in the US) and a third-party transcriber who will have signed appropriate confidentiality and data sharing agreements before any data are shared. | | |
| 14. I confirm that I am an Oxford University student currently living in the UK, and that I am 18-25 years old. | | |
| 15. I consent to be contacted via SMS to complete weekly surveys online during Trinity Term 2022, and to fill in a short follow-up survey at the end of the term. | | |
| 16. (Optional) I agree that the research team may retain my contact details so that I may be contacted in the future by the research team to invite me to participate in future studies of a similar nature. | | |
| Name of Participant | Date | Signature |
| Name of Researcher | Date | <br>Signature |